CLINICAL TRIAL: NCT07250698
Title: Postprandial Walks for Glucose Control in Type 2 Diabetes in Pregnancy
Brief Title: Glucose Control in Type 2 Diabetes in Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Marwan Ma'ayeh, Assistant Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-06-FB-0155
Record Dates: First submitted 2025-09-24; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pregestational Diabetes; Type 2 Diabetes
Keywords: exercise; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-prandial walk (Active Comparator): Participants in this arm of the study will be instructed to walk for 20 minutes after each meal (breakfast, lunch, and dinner). They will also be given a continuous glucose monitor and a FitBit, to wear throughout their participation in the study.
  Interventions: Behavioral: Exercise
- Standard of Care (No Intervention): Participants in this arm will be given the regular counseling on the importance of exercise during pregnancy, but not instructed to walk after each meal. They will receive a continuous glucose monitor and FitBit to wear throughout their participation in the study.

INTERVENTIONS:
Behavioral: Exercise — This intervention consists of instructions to walk for 20 minutes after each meal.
  Arms: Post-prandial walk

SUMMARY:
The goal of this clinical trial is to evaluate the effect of physical activity on glucose control in pregnant patients with pregestational Type 2 diabetes. The main question it seeks to answer is "will physical activity following a meal improve blood sugar control in pregnant women with Type 2 diabetes?" Researchers will compare the glucose control of two groups: one that walks for 20 minutes after each meal, and one that does not.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Known diagnosis of Type 2 diabetes OR meets new diagnosis of Type 2 diabetes in the first trimester (up to 13 weeks and 6 days)
* Age ≥18 and <50 years
* Gestational age <32 weeks 0 days gestation

Exclusion Criteria:

* Non-English as the primary language
* Inability to participate in 20 minutes of walking at a time
* Known or suspected fetal anomaly or aneuploidy
* Prisoners
* Management of diabetes outside of study location

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Time in Range | Between 34 and 36 weeks gestation.
  Our primary outcome is the time in range (via CGM data) during the management of Type 2 diabetes in pregnancy between 34 and 36 weeks gestation.

SECONDARY OUTCOMES:
Duration of postprandial walk | From enrollment to delivery, an average of 6 months
  Duration of postprandial walk (in minutes)
Sleep duration | From enrollment to delivery, an average of 6 months
  Amount of time spent sleeping
Baseline heart rate | From enrollment to delivery, an average of 6 months
  Heart rate when not exercising
Maximal heart rate during walks | From enrollment to delivery, an average of 6 months
  Maximal heart rate during postprandial walks
Frequency of aerobic exercise per week | From enrollment to delivery, an average of 6 months
  Number of times a participant engages in aerobic exercise each week
Mean glucose level | From enrollment to delivery, an average of 6 months
  Average blood sugar level
Blood Glucose Excursions | From enrollment to delivery, an average of 6 months
  Changes in blood glucose
Fasting blood sugar | From enrollment to delivery, an average of 6 months
  Blood sugar following a fast
Total daily insulin dose | From enrollment to delivery, an average of 6 months
  The total amount of insulin administered to the participant daily
Rates of fetal demise | From enrollment to delivery, an average of 6 months
  Whether fetal death occurs prior to delivery
Rates of fetal growth restriction among participants | From enrollment to delivery, an average of 6 months
  When the fetus is considered small for gestational age at any point in pregnancy
Rates of preeclampsia among participants | From enrollment to delivery, an average of 6 months
  Occurrence of preeclampsia during pregnancy
Rates of placental abruption among participants | From enrollment to delivery, an average of 6 months
Mode of delivery | From enrollment to delivery, an average of 6 months
  Cesarean or vaginal
Number of participants with indication for cesarean delivery | From enrollment to delivery, an average of 6 months
Presence of shoulder dystocia | Duration of delivery, up to 72 hours
  Vaginal deliveries
Quantitative blood loss | From onset of labor to hospital discharge, up to 42 days post-delivery
  mL
Postpartum hemorrhage | From delivery to hospital discharge, up to 42 days post-delivery
  Defined as quantitative blood loss >1000 mL
Occurrence of Infection | From delivery to hospital discharge, up to 42 days
  Chorioamnionitis or postpartum endometritis prior to discharge
Neonatal birth weight | From delivery to hospital discharge, up to 42 days
  Grams
APGAR Scores | From delivery to hospital discharge, up to 1 year
  Scored from 0-10, with 10 being the best outcome
Incidence of Neonatal Infection | From delivery to hospital discharge, up to 1 year
  Sepsis, fever, positive cultures, or a suspicious clinical course that warrants antibiotics treatment
Rates of respiratory distress syndrome amongst participant infants | From delivery to hospital discharge, up to 1 year
Rates of necrotizing enterocolitis amongst participant infants | From delivery to hospital discharge, up to 1 year
Rates Neonatal Intensive Care Unit admission amongst participant infants | From deliver to NICU admission, up to 1 year
Days in the NICU | From NICU admission to NICU discharge, up to 1 year
Hemoglobin A1c | At time of randomization, up to 32 weeks gestation
  Blood Hemoglobin A1c level
Hemoglobin A1c | Between 34 and 36 weeks gestation
  Blood Hemoglobin A1c levels
C-peptide | Collected at time of randomization, up to 32 weeks gestation
  Blood c-peptide levels
C-peptide | Between 34 and 36 weeks gestation
  Blood c-peptide levels
Insulin | At time of randomization, up to 32 weeks gestation
  Blood insulin levels
Insulin | Between 34 and 36 weeks gestation
  Blood insulin level
Leptin | At time of randomization, up to 32 weeks gestation
  Blood leptin level
Leptin | Between 34 and 36 weeks gestation
  Blood leptin level
Adipoleptin | At time of randomization, up to 32 weeks gestation
  Blood adipoleptin
Adipoleptin | Between 34 and 36 weeks gestation
  Blood adipoleptin level
Body fat mass | At time of randomization, up to 32 weeks gestation
  Mass of body fat determined using bioelectrical impedance analysis
Body fat mass | Between 34 and 36 weeks gestation
  Mass of body fat determined using bioelectrical impedance analysis
Body fat percentage | At time of randomization, up to 32 weeks gestation
  Body fat percentage determined via bioelectrical impedance analysis
Body fat percentage | Between 34 and 36 weeks gestation
  Body fat percentage determined via bioelectrical impedance analysis
Fat free mass | Time of randomization, up to 32 weeks
  Measure of body composition, determined by bioelectrical impedance analysis
Fat free mass | Between 34 and 36 weeks gestation
  Measure of body composition, determined by bioelectrical impedance analysis
Total body water | At time of randomization, up to 32 weeks gestation
  Amount of water in the body, determined by bioelectrical impedance analysis
Total body water | Between 34 and 36 weeks gestation
  Amount of water in the body, determined by bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virginia Medical School, Macon and Joan Brock Virginia Health Sciences at Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Colberg SR, Zarrabi L, Bennington L, Nakave A, Thomas Somma C, Swain DP, Sechrist SR. Postprandial walking is better for lowering the glycemic effect of dinner than pre-dinner exercise in type 2 diabetic individuals. J Am Med Dir Assoc. 2009 Jul;10(6):394-7. doi: 10.1016/j.jamda.2009.03.015. Epub 2009 May 21. PMID 19560716
- [Background] Christie HE, Chang CR, Jardine IR, Francois ME. Three short postmeal walks as an alternate therapy to continuous walking for women with gestational diabetes. Appl Physiol Nutr Metab. 2022 Oct 1;47(10):1031-1037. doi: 10.1139/apnm-2021-0619. Epub 2022 Aug 19. PMID 35985050
- [Background] Andersen MB, Fuglsang J, Ostenfeld EB, Poulsen CW, Daugaard M, Ovesen PG. Postprandial interval walking-effect on blood glucose in pregnant women with gestational diabetes. Am J Obstet Gynecol MFM. 2021 Nov;3(6):100440. doi: 10.1016/j.ajogmf.2021.100440. Epub 2021 Jun 30. PMID 34216833
- [Background] Jovanovic-Peterson L, Durak EP, Peterson CM. Randomized trial of diet versus diet plus cardiovascular conditioning on glucose levels in gestational diabetes. Am J Obstet Gynecol. 1989 Aug;161(2):415-9. doi: 10.1016/0002-9378(89)90534-6. PMID 2764059
- [Background] Garcia-Patterson A, Martin E, Ubeda J, Maria MA, de Leiva A, Corcoy R. Evaluation of light exercise in the treatment of gestational diabetes. Diabetes Care. 2001 Nov;24(11):2006-7. doi: 10.2337/diacare.24.11.2006. No abstract available. PMID 11679479
- [Background] Fishel Bartal M, Ashby Cornthwaite JA, Ghafir D, Ward C, Ortiz G, Louis A, Cornthwaite J, Chauhan SSP, Sibai BM. Time in Range and Pregnancy Outcomes in People with Diabetes Using Continuous Glucose Monitoring. Am J Perinatol. 2023 Apr;40(5):461-466. doi: 10.1055/a-1904-9279. Epub 2022 Jul 20. PMID 35858653
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693
- [Background] Gregory ECW, Ely DM. Trends and Characteristics in Prepregnancy Diabetes: United States, 2016-2021. Natl Vital Stat Rep. 2023 May;72(6):1-13. PMID 37256333

DOCUMENTS (3):
  • Study Protocol (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT07250698/Prot_000.pdf
  • Informed Consent Form: Experimental Consent Form (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT07250698/ICF_001.pdf
  • Informed Consent Form: Control Consent Form (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT07250698/ICF_002.pdf